CLINICAL TRIAL: NCT04230564
Title: Characteristics, Treatment Patterns, and Clinical Outcomes in Non-intensive Chemotherapy Acute Myeloid Leukemia (AML) Patients - a US Real-World Study Using Electronic Medical Record Data
Brief Title: Acute Myeloid Leukemia Real World Treatment Patterns
Status: Withdrawn | Type: Observational
Why Stopped: Study was cancelled prior to any enrollment
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1371038
Record Dates: First submitted 2020-01-13; First posted 2020-01-18 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2021-02

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: Acute Myeloid Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; venetoclax; glasdegib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- AML: Patients diagnosed with AML
  Interventions: Drug: azacitidine; Drug: venetoclax; Drug: glasdegib

INTERVENTIONS:
Drug: azacitidine — Patients taking azacitidine
Drug: venetoclax — patients taking venetoclax
Drug: glasdegib — patients taking glasdegib

SUMMARY:
Among patients with a diagnosis of AML who received non-intensive chemotherapy:

* Describe patient demographic and clinical characteristics
* Describe treatment patterns
* Describe effectiveness outcomes
* Evaluate tumor response

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

1. Confirmed diagnosis of AML on or after 01 January 2012 through Clinical Research Nurse (CRN) review of provider documentation of AML diagnosis in the medical record.
2. Receipt of non-intensive therapy at any point during first line therapy following initial AML diagnosis. For this study, non-intensive therapy will be defined as 1 of the following agents, alone or in combination with any other agent:

   1. AZA
   2. GLAS
   3. VEN
3. Age ≥18 years at initial diagnosis of AML.

Exclusion Criteria:

Patients meeting any of the following criteria will not be included in the study:

1. Record of 1 or more of the following confounding diagnoses at any point before or after AML diagnosis: Acute lymphoblastic leukemia; acute promyelocytic leukemia, aggressive systemic mastocytosis; hypereosinophilic syndrome and/or chronic eosinophilic leukemia; dermatofibrosarcoma protuberans; gastrointestinal stromal tumors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include adult patients diagnosed with AML who, at any point during first line therapy, received non-intensive therapy
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-10-31 (Estimated); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | January 1, 2012 to January 10, 2020
  Overall survival was the duration from diagnosis of disease to death.
Event Free Survival | January 1, 2012 to January 10, 2020
  Time from the treatment initiation date to the date of treatment failure (TF), relapse from CR or better, or death from any cause, whichever comes first
Relapse Free Survival | January 1, 2012 to January 10, 2020
  Time from the treatment initiation date to the date of a relapse event, or death from any cause, whichever comes first
Best response | January 1, 2012 to January 10, 2020
  Best response recorded from treatment start until disease progression/recurrence
Time to best response | January 1, 2012 to January 10, 2020
  Time from treatment initiation until best response recorded
Duration of best response | January 1, 2012 to January 10, 2020
  Time from best response achieved until lose of response or the end of the record, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.